CLINICAL TRIAL: NCT00892879
Title: A Randomized Trial of Single Port Laparoscopic Cholecystectomy Versus Four Port Laparoscopic Cholecystectomy
Brief Title: A Trial of Single Port Laparoscopic Cholecystectomy Versus Four Port Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Paul Hansen, MD, Providence Health & Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHS IRB # 09-14A
Record Dates: First submitted 2009-04-27; First posted 2009-05-05 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single port laparoscopic device
  Interventions: Device: Laparoscopic cholecystectomy surgery
- 2 (Active Comparator): Four-port laparoscopic device
  Interventions: Device: Laparoscopic cholecystectomy surgery

INTERVENTIONS:
Device: Laparoscopic cholecystectomy surgery — Single port laparoscopic cholecystectomy surgery versus a standard four port device.
  Other Names: ACS Triport, Advanced Surgical Concepts, Ireland

SUMMARY:
This is a single-institution, prospective, one-to-one randomized controlled research study. Subjects medically determined to need a cholecystectomy will be consented for surgery and study participation prior to enrolment in this study. Patients will then be randomized to receive either a single port laparoscopic cholecystectomy or a four port laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative diagnosis of one of the following:

  * Pancreatic cholecystitis
  * Biliary cholic
  * Biliary dyskinesia
  * Choledocholithiasis status post endoscopic retrograde cholangiopancreatography/sphincterotomy
  * Gallbladder polyps
  * Other diagnosis at the discretion of the surgeon

Exclusion Criteria:

* Acute cholecystitis
* Gallstones > 2.5cm in length on ultrasound
* Suspected presence of common duct stones
* History of jaundice
* History of gallstone pancreatic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Post-operative pain scores (visual analogue pain scale from 0-10)assessed on post-operative day 1 and at the post-operative follow up visit in clinic. The mean pain scores will be compared using student's t-test. | 3-6 weeks

SECONDARY OUTCOMES:
The postoperative infection rate will be monitored and compared for patients undergoing single port laparoscopic cholecystectomy and four port laparoscopic cholecystectomy. | 3-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Hansen, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

REFERENCES:
- [Derived] Ma J, Cassera MA, Spaun GO, Hammill CW, Hansen PD, Aliabadi-Wahle S. Randomized controlled trial comparing single-port laparoscopic cholecystectomy and four-port laparoscopic cholecystectomy. Ann Surg. 2011 Jul;254(1):22-7. doi: 10.1097/SLA.0b013e3182192f89. PMID 21494123